CLINICAL TRIAL: NCT06918769
Title: The Application of a Novel Urinalysis System (UF-5000) for Reducing Unnecessary Antibiotic Use in Clinical Suspected UTI Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Sysmex Asia Pacific (Industry)
Responsible Party: Principal Investigator, Yung NA, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HKURO202201
Record Dates: First submitted 2024-05-07; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Urinary Tract Infections; Urinary Tract Infection Lower Acute
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Active Comparator): Empirical antibiotics without bacterial information
  Interventions: Drug: Empirical antibiotics
- Experimental Arm (Experimental): Antibiotics prescription with reference from study device. High bacterial count suggests likelihood of active UTI and indicated for antibiotics treatment; while low bacterial count suggests UTI not likely and antibiotics treatment will be delayed until urinary culture result confirms ongoing UTI.
  Interventions: Diagnostic Test: Sysmex UF-5000 system

INTERVENTIONS:
Diagnostic Test: Sysmex UF-5000 system — Provide real time bacterial count in urine samples and Gram-staining results. High bacterial count suggests likelihood of active UTI and indicated for antibiotics treatment; while low bacterial count suggests UTI not likely.
  Arms: Experimental Arm
Drug: Empirical antibiotics — Empirical antibiotics per local guideline/ investigator's discretion for urinary tract infection
  Arms: Control Arm

SUMMARY:
Urinary tract infection (UTI) is one of the most common diseases in population while antibiotic resistant in UTI has become a critical problem in Hong Kong, that a large proportion of the bacteria in UTI resistant to commonly used anti-UTI antibiotic treatment. This is largely due to the empirical treatment (i.e. no bacteria information is available at the time of treatment) and overtreatment of antibiotics in the past decades. Some patients who did not actually have UTI were prescribed with antibiotics because they have symptoms similar to UTI.

In order to avoid unnecessary use of antibiotics and therefore reduce the antibiotic resistance rates of UTI, we propose to apply a new urine sediment analyzer (UF-5000) in clinical practice for UTI which could provide quick label for potential bacteria in urine, and give more information on the possible species of the bacteria.

UF-5000 is a urine sediment analyzer manufactured by Sysmex Ltd. (Japan), it is widely used in central laboratories of hospitals and private laboratories, but not commonly seen in out-patient clinic setting. UF-5000 is capable of counting the amount of bacteria present in the given urine sample and provide Gram staining*, with results available within 5 minutes. While routine urine culture would take around 3 days.

A study done by The University of Hong Kong in 2019 has shown that UF-5000 has higher accuracy than conventional dipstick, with reliable Gram staining result. It has a negative-prediction value of 96%, which means it could accurately identify the cases who had no UTI but only similar symptoms. Those cases were mostly inflammatory diseases that did not require antibiotics.

This study aims to evaluate whether bacteria information provided by UF-5000 would be able to guide a precision use of antibiotic treatment and avoid unnecessary antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients who are suspected to have LUTs in outpatient clinic.
2. Willing to consent to participate the trial.
3. Be able to understand the nature of the study.

Exclusion Criteria:

1. Any suspected or known sexual transmitted diseases. (Such as gonorrhea, etc.)
2. Use of any systematic antibiotics or antiviral treatment within two weeks
3. With evidence of systematic infection including high fever, significantly increase of blood white blood cell count, etc.
4. Known or suspected allergic history/adverse drug reactions to any antibiotics
5. With previous history of multidrug resistant (MDR) bacterial infection.
6. Any medical history that indicates the need of immediate antibiotics treatment, such as chronic conditions and/or taking immunosuppressants.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects assigned with "Delay antibiotics treatment" in the intervention group that has confirmed no clinical indication for antibiotics treatment | 1 week
  The rate of unnecessary antibiotics use avoided in the intervention group. Defined as proportion of subjects assigned with "Delay antibiotics treatment" as indicated by low real-time bacterial count in urine that had negative or clinically insignificant urine culture result in one week

SECONDARY OUTCOMES:
Number of subjects achieved urinary sterility after antibiotics treatment in confirmatory urine test | 1 week
  Defined as negative white blood cell in urine dipstick and no growth in urine culture. Only applies to subjects that have finished a course of antibiotics treatment under study setting.
Number of participants that persist to have baseline lower tract urinary symptoms as assessed in CTCAE 4.0 | 1 week
  The symptoms would be assessed through phone follow-up.
Number of participants with antibiotics treatment-related adverse events as assessed by CTCAE v4.0 | 2 weeks
  The symptoms would be assessed through phone follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No